CLINICAL TRIAL: NCT00570492
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Evaluate the Effects of a One-Year Course of Fluticasone Furoate Nasal Spray 110mcg QD on Growth in Pre-Pubescent, Pediatric Subjects With Perennial Allergic Rhinitis
Brief Title: Phase 4 Fluticasone Furoate Nasal Spray (VERAMYST) Long Term Pediatric Growth Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FFR101782
Record Dates: First submitted 2007-12-06; First posted 2007-12-11 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: allergic rhinitis; fluticasone furoate nasal spray; growth
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray
- Fluticasone furoate nasal spray (Experimental)
  Interventions: Drug: Fluticasone furoate nasal spray

INTERVENTIONS:
Drug: Fluticasone furoate nasal spray — Fluticasone furoate nasal spray 110mg QD
  Arms: Fluticasone furoate nasal spray
Drug: Placebo nasal spray — Placebo nasal spray
  Arms: Placebo nasal spray

SUMMARY:
The primary objective of this study is to characterize, as accurately as possible, the estimation of the difference in pre-pubescent growth velocities between subjects treated continuously for one year with FFNS 110mcg QD, the highest dose approved for pediatric use in the US, and placebo nasal spray as determined by stadiometry.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated informed consent obtained from the subject's legal parent/guardian. Adequate provisions for assent of children should be provided in accordance with the IRB and any local governance.
* Age: 5 to less than 7.5 years for females and 5 to less than 8.5 years for males at Visit 1.
* Subjects must have a diagnosis and history of perennial allergic rhinitis (PAR) as follows:
* At least a one year clinical history and treatment of PAR (written or verbal confirmation from the treating physician) and,
* A documented, positive skin test to an appropriate perennial allergen (animal dander, house dust mites, cockroaches and/or mold) or documented, historical, in vitro test results for a specific IgE (such as RAST, PRIST) within the past 12 months prior to Visit 1 will be allowed. A positive skin test during Visit 1 will also be allowed. A positive skin test is defined as a wheal 3mm larger than the diluent control for prick testing.

Note: Subjects who meet the above criteria and who may also have seasonal allergic rhinitis (SAR) and/or non-allergic rhinitis (NAR) are eligible for randomization.

* At Visit 2, the daily rTNSS on any 4 of the last 7 days prior to Visit 2 must be 5. Subjects should refrain from using rescue medication during the 7 days prior to Visit 2.
* Pre-pubescence: Tanner Staging equal to 1 for all classifications as assessed by the investigator during each of the five baseline study visits (Visit 1 through Visit 5). The same investigator should perform this assessment throughout the study for a respective subject, if possible, for consistency of assessment. Details are provided in the SPM.
* Current height measurement via standardized stadiometer is within the 3rd and 97th percentile according to the CDC and any local longitudinal standard height charts for age and gender as provided in the SPM (Visit 1 through Visit 5).
* Body weight and body mass index between the 3rd and 97th percentile according to the US CDC standards and any local standards as assessed during each of the five baseline study visits (Visit 1 through Visit 5). The US CDC standards are provided in the SPM.
* Compliance: Subject's parent/guardian is literate and both subject and parent/guardian are deemed capable of complying with all study procedures to include proper study drug administration, daily e-diary completion, in-clinic laboratory assessments, and in-home 24 hour urine collection during the 76 weeks of study participation (Visit 1 through Visit 5).

Exclusion criteria:

* A history or evidence of abnormal growth. Any previous or current condition that affects growth, including sleep disorders.
* Asthma, with the exception of mild intermittent asthma [National Asthma Education and Prevention Program, 2007] (Note: Subjects will be allowed to use short-acting inhaled beta2 agonists only on an as needed basis.)
* A history of nasal or sinus surgery, septal perforation, or severe obstruction in the nose (e.g. nasal polyps).
* Any other significant concomitant medical condition. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study. (Visit 1 through Visit 5)
* Any prior or current use of any medication/treatment that might affect growth including, but not limited to, methylphenidate hydrochloride, thyroid hormone, growth hormone, anabolic steroids, calcitonin, estrogens, progestins, biphosphonates, anticonvulsants or phosphate binding antacids. (Visit 1 through Visit 5).
* Use of corticosteroids, defined as:
* Inhaled, intranasal, or high potency topical (to include dermatological, optic and otic) corticosteroids within 6 weeks prior to Visit 1 or during the baseline period (Visit 1 through Visit 5).
* Systemic corticosteroids (to include oral and injectable) within 12 weeks prior to Visit 1 or during the baseline period (Visit 1 through Visit 5).
* Use of other allergy medications within an appropriate timeframe relative to Visit 1 to allow the medication to be eliminated or no longer producing an effect as well as during the baseline period (Visit 1 through Visit 5) including, but not limited to:
* Intranasal cromolyn - 14 days
* Short-acting prescription and OTC antihistamines - 3 days
* Long acting (second-generation) antihistamines (other than the loratadine syrup supplied by GSK to treat uncontrolled symptoms of PAR) including fexofenadine, cetirizine, desloratadine, and astemizole - 10 days
* Long-acting antihistamine: astemizole - 12 weeks
* Intranasal antihistamines (e.g. azelastine) -2 weeks
* Oral or intranasal decongestants - 3 days
* Intranasal, oral or inhaled anticholinergics - 3 days
* Oral antileukotrienes - 3 days
* Subcutaneous omalizumab - 5 months
* Immunotherapy initiated or adjusted within 30 days prior to Visit 1 or during the baseline period (Visit 1 through Visit 5) noting that no significant changes in the dose, concentration or dilution will be allowed during the study.
* Use of immunosuppressive medications 8 weeks prior to screening or during the baseline period (Visit 1 through Visit 5) of the study.
* Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole. (Visit 1 through Visit 5)
* Allergy/Intolerance
* Known hypersensitivity to corticosteroids or any excipients in the nasal spray
* Known hypersensitivity to the antihistamine or decongestant being provided for worsening symptoms of rhinitis during the conduct of the study.
* Exposure to varicella (Chickenpox) or measles during the 3 weeks prior to screening or during the baseline period (Visit 1 through Visit 5), if non-immune. A diagnosis of varicella or measles during the baseline period is exclusionary as well.
* Recent exposure to an investigational study drug within 30 days prior toVisit 1.
* Affiliation with investigational site.
* Findings of a clinically significant, abnormal screening (Visit 1) clinical laboratory test.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 474 (Actual)
Dates: Start 2007-11-26; Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (43):
  - GSK Investigational Site, Oxford, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Richmond, Virginia
- Argentina (5):
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Santa Fe
- Canada (7):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- France (3):
  - GSK Investigational Site, Laon
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Montpellier
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria
- GSK Investigational Site, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lee LA, Sterling R, Maspero J, Clements D, Ellsworth A, Pedersen S. Growth velocity reduced with once-daily fluticasone furoate nasal spray in prepubescent children with perennial allergic rhinitis. J Allergy Clin Immunol Pract. 2014 Jul-Aug;2(4):421-7. doi: 10.1016/j.jaip.2014.04.008. Epub 2014 May 21. PMID 25017530
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR101782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening and a 16-week Baseline Period (Pd.), participants (par.) were randomized 1:1 to each treatment arm during the 52-week Treatment Pd. After the Treatment Pd., par. entered an 8-week Follow-up (FU) Pd. during which all par. received placebo nasal spray. Par. completing at least 12 weeks of treatment were to complete the FU Pd.
Groups:
- Placebo: Baseline Period: Placebo nasal spray administered once daily (OD) as 2 sprays per nostril to all enrolled participants during the 16-week Single-blind Baseline period, to assess the baseline growth velocity
- Placebo: Double-blind Treatment Period: Participants were randomized to receive matching placebo nasal spray OD as 2 sprays per nostril during the 52-week Double-blind Treatment Period
- FFNS 110 mcg: Double-blind Treatment Period: Participants were randomized to receive fluticasone furoate nasal spray (FFNS) 110 micrograms (mcg) OD as 2 sprays per nostril during the 52-week Double-blind Treatment Period
Period: 16-week Single-blind Baseline Period
Arm/Group | Placebo: Baseline Period | Placebo: Double-blind Treatment Period | FFNS 110 mcg: Double-blind Treatment Period
Started | 910 | 0 | 0
Completed | 474 | 0 | 0
Not Completed | 436 | 0 | 0
Not completed — Didn't Meet Inclusion/Exclusion Criteria | 98 | 0 | 0
Not completed — Didn't Meet Randomization Criteria | 263 | 0 | 0
Not completed — Withdrawal by Subject | 56 | 0 | 0
Not completed — Protocol Violation | 15 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Randomized but Did'nt Receive Treatment | 1 | 0 | 0
Period: 52-week Double-blind Treatment Period
Arm/Group | Placebo: Baseline Period | Placebo: Double-blind Treatment Period | FFNS 110 mcg: Double-blind Treatment Period
Started | 0 | 237 | 237
Completed | 0 | 187 | 186
Not Completed | 0 | 50 | 51
Not completed — Withdrawal by Subject | 0 | 20 | 20
Not completed — Protocol Violation | 0 | 12 | 15
Not completed — Lost to Follow-up | 0 | 5 | 7
Not completed — Adverse Event | 0 | 5 | 5
Not completed — Physician Decision | 0 | 2 | 4
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Reached Protocol-defined Stop Criteria | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo nasal spray OD (as 2 sprays per nostril at each time point) in the 16-week Single-blind Baseline Period, in the following 52-week Double-blind Treatment Period (after randomization), and then in the 8-week Single-blind Follow-up Period.
- FFNS 110 mcg: Participants received placebo nasal spray OD (as 2 sprays per nostril at each time point) in the 16-week Single-blind Baseline Period, and then received FFNS 110 mcg OD in the following 52-week Double-blind Treatment Period. Participants again received placebo nasal spray OD in the 8-week Single-blind Follow-up Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | FFNS 110 mcg | Total
Number analyzed (Participants) | 237 | 237 | 474
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all participants who had been randomized to and received at least one dose of Double-blind study medication.
  Years | 6.61 (0.969) | 6.64 (0.933) | 6.63 (0.950)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all participants who had been randomized to and received at least one dose of Double-blind study medication.
  Participants
    Female | 73 | 75 | 148
    Male | 164 | 162 | 326
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all participants who had been randomized to and received at least one dose of Double-blind study medication.
  participants
    African American (Amc)/African Heritage | 16 | 12 | 28
    Amc Indian or Alaska Native (Alk N) | 19 | 18 | 37
    Asian | 7 | 5 | 12
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    White | 189 | 199 | 388
    African Amc/African and Amc Indian or Alk N | 1 | 0 | 1
    African Amc/African Heritage and White | 1 | 2 | 3
    Amc Indian or Alk N and White | 1 | 0 | 1
    Asian and White | 1 | 1 | 2
    Native Hawaiian/ Other Pacific Islander and White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Growth Velocity of Pre-pubescent Pediatric Participants to the End of the 52-week Double-blind (DB) Treatment Period
Description: Height was measured (triplicate measurements) in pre-pubescent pediatric participants via stadiometry at each clinic visit during the entire 76-week study period (16-week Baseline Period, 52-week DB Treatment Period and 8-week Follow-up Period). Growth velocity was calculated by fitting a regression line to all height measurements recorded for the participant during the period and was determined by the slope of the fitted regression line. Change from Baseline was calculated as the value over the 52-week Treatment Period minus the value over the 16-week Baseline Period.
Time Frame: Baseline Period (Weeks -16 to 0) and DB Treatment Period (Weeks 1 to 52)
Population: Growth Population: all randomized participants with height assessments via stadiometry from at least three post-randomization clinic visits during the DB Treatment Period
Measure: Least Squares Mean (Standard Error); unit: Centimeters per year (cm/year)
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 218 | 217
Centimeters per year (cm/year) | 5.46 (0.10) | 5.19 (0.10)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.270, 95% CI 2-sided [-0.48 to -0.06] — An analysis of covariance (ANCOVA) was performed to estimate the mean treatment difference in growth velocity over the treatment period, adjusting for baseline growth velocity, age, gender, and country

2. Secondary Outcome: Mean 24-hour Urinary Free Cortisol Excretion
Description: Hypothalamic-pitiutary-adrenal (HPA) axis function was assessed by the measurement of urinary free cortisol, using urine samples collected over the course of 24 hours by the parent/guardian in the participants' home on an out-patient basis within 7 days prior to the indicated time points. Detailed verbal instructions and a take-home instruction card on how to conduct the 24-hour urine collection were provided to the parent/guardian before each collection interval.
Time Frame: Randomization/end of 16-week Baseline Period (Week 0), End of 52-week DB Treatment Period (Week 52), and end of 8-week Follow-up Period (Week 60)
Population: Urine Cortisol Population: all randomized participants excluding those whose urine samples were considered to have confounding factors affecting the interpretation of the 24-hour urinary cortisol results. One participant in each arm had a Baseline value <1.0 and was not analyzed. Some participants had samples that were not acceptable for analysis.
Measure: Mean (Standard Deviation); unit: Micrograms per 24 hours (mcg/24 hours)
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 168 | 172
Micrograms per 24 hours (mcg/24 hours)
  End of 16-week Baseline Period, n=168, 172 | 9.771 (6.0479) | 9.242 (5.5821)
  End of 52-week DB Treatment Period, n=163, 169 | 11.340 (9.6775) | 11.125 (9.2195)
  End of 8-week Follow-up Period, n=161, 167 | 10.615 (6.6903) | 10.311 (5.9986)

3. Secondary Outcome: Number of Participants With the Indicated Shifts From Baseline in Nasal Examination (NE) Results
Description: NE included the evaluation of the size of ulcers/polyps (of nasal turbinates/septa) and assessment for mucosal bleeding (MB) at all study visits. Polyps are non-cancerous growths; ulcers are breaks in the skin/mucous membrane with loss of surface tissue, disintegration, and necrosis of epithelial tissue. For MB, Improved=shift from present (>=1 nostril) to absent (both nostrils); Worsened=shift from absent (both nostrils) to present (>=1 nostril). For polyps/ulcers, Improved=shift from large to small or from small to none; Worsened=shift from none to small or from small to none (>=1 nostril).
Time Frame: Baseline Period (Weeks -16 to 0) and DB Treatment Period (Weeks 1 to 52)
Population: Intent-to-Treat (ITT) Population: all participants who had been randomized to and received at least one dose of double-blind study medication. Most participants received examinations at each visit; however, on some occasions, some assessments were not completed for various reasons.
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 191 | 188
participants
  Mucosal Bleeding, Improved | 1 | 0
  Mucosal Bleeding, No Change | 190 | 187
  Mucosal Bleeding, Worsened | 0 | 1
  Ulcers, Improved | 0 | 0
  Ulcers, No Change | 191 | 188
  Ulcers, Worsened | 0 | 0
  Polyps, Improved | 1 | 0
  Polyps, No Change | 190 | 188
  Polyps, Worsened | 0 | 0

4. Secondary Outcome: Mean Values for the Laboratory Parameters of Alkaline (Alk) Phosphatase (P), Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST)
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: Alk P, ALT, and AST.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: ITT Population. Only those participants remaining in the study and contributing viable samples at the various time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 234
International Units per liter (IU/L)
  Alk P, Baseline Period, n=231, 234 | 246.8 (57.45) | 249.8 (67.81)
  Alk P, DB Treatment Period, n=184, 182 | 261.9 (61.96) | 262.9 (71.22)
  Alk P, Follow-up Period, n=175, 174 | 264.2 (59.67) | 264.6 (67.44)
  ALT, Baseline Period, n=231, 234 | 14.8 (4.54) | 15.1 (4.73)
  ALT, DB Treatment Period, n=184, 182 | 15.9 (8.50) | 15.8 (5.12)
  ALT, Follow-up Period, n=175, 174 | 16.7 (14.41) | 17.2 (13.15)
  AST, Baseline Period, n=229, 232 | 27.4 (4.89) | 28.1 (4.89)
  AST, DB Treatment Period, n=175, 179 | 27.0 (5.49) | 27.6 (4.87)
  AST, Follow-up Period, n=169, 174 | 27.7 (8.93) | 28.3 (10.44)

5. Secondary Outcome: Mean Values for the Laboratory Parameters if Albumin and Total Protein
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: Albumin and Total Protein.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 234
Grams per liter (g/L)
  Albumin, Baseline Period, n=231, 234 | 45.8 (2.29) | 46.0 (2.33)
  Albumin, DB Treatment Period, n=184, 182 | 45.7 (2.24) | 45.9 (2.25)
  Albumin, Follow-up Period, n=175, 175 | 45.8 (2.31) | 45.6 (2.36)
  Total Protein, Baseline Period, n=231, 234 | 72.0 (3.78) | 71.9 (4.30)
  Total Protein, DB Treatment Period, n=184, 182 | 71.7 (3.76) | 71.7 (3.95)
  Total Protein, Follow-up Period, n=175, 175 | 71.5 (3.66) | 71.5 (3.83)

6. Secondary Outcome: Mean Values for the Laboratory Parameters of Total Bilirubin and Creatinine
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: Total Bilirubin and Creatinine.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Micromoles (µmol)/L
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 234
Micromoles (µmol)/L
  Total Bilirubin, Baseline Period, n=231, 234 | 6.9 (2.43) | 7.2 (3.40)
  Total Bilirubin, DB Treatment Period, n=184, 182 | 7.2 (2.69) | 7.7 (3.56)
  Total Bilirubin, Follow-up Period, n=175, 175 | 7.0 (2.72) | 7.1 (3.14)
  Creatinine, Baseline Period, n=231, 234 | 43.3 (7.98) | 43.6 (7.96)
  Creatinine, DB Treatment Period, n=184, 182 | 45.0 (8.34) | 44.6 (8.16)
  Creatinine, Follow-up Period, n=175, 175 | 44.5 (7.38) | 45.0 (7.72)

7. Secondary Outcome: Mean Values for the Laboratory Parameters of Glucose, Calcium, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN)
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: Glucose, Calcium, Potassium, Sodium, and Urea/BUN.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/L
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 234
Millimoles (mmol)/L
  Glucose, Baseline Period, n=230, 231 | 4.83 (0.683) | 4.86 (0.690)
  Glucose, DB Treatment Period, n=184, 182 | 4.82 (0.782) | 4.78 (0.720)
  Glucose, Follow-up Period, n=175, 175 | 4.87 (0.840) | 4.85 (0.700)
  Calcium, Baseline Period, n=229, 232 | 2.441 (0.0786) | 2.435 (0.0993)
  Calcium, DB Treatment Period, n=175, 179 | 2.437 (0.0776) | 2.440 (0.0847)
  Calcium, Follow-up Period, n=169, 173 | 2.438 (0.0769) | 2.436 (0.0820)
  Potassium, Baseline Period, n=229, 232 | 4.30 (0.404) | 4.31 (0.437)
  Potassium, DB Treatment Period, n=175, 179 | 4.30 (0.373) | 4.30 (0.345)
  Potassium, Follow-up Period, n=169, 173 | 4.28 (0.362) | 4.32 (0.409)
  Sodium, Baseline Period, n=231, 234 | 139.4 (1.90) | 139.3 (1.83)
  Sodium, DB Treatment Period, n=184, 182 | 139.1 (1.65) | 139.2 (1.58)
  Sodium, Follow-up Period, n=175, 175 | 139.3 (1.89) | 139.4 (2.19)
  Urea/BUN, Baseline Period, n=231, 235 | 4.99 (1.897) | 4.77 (1.195)
  Urea/BUN, DB Treatment Period, n=184, 182 | 4.82 (1.315) | 4.82 (1.294)
  Urea/BUN, Follow-up Period, n=175, 175 | 4.93 (1.219) | 4.75 (1.274)

8. Secondary Outcome: Mean Hematology Values for Basophil, Eosinophil, Lymphocyte, White Blood Cell (WBC), Monocyte, Segmented Neutrophil (Neu), and Platelet Counts
Description: Participants in the study were evaluated for the following hematology laboratory parameters at the indicated time points: Basophil, Eosinophil, Lymphocyte, White Blood Cell (WBC), Monocyte, Segmented Neutrophil (Neu), and Platelet counts.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells (Gi)/L
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 228 | 231
Giga (10^9) cells (Gi)/L
  Basophil, Baseline Period, n=228, 231 | 0.026 (0.0176) | 0.025 (0.0151)
  Basophil, DB Treatment Period, n=186, 188 | 0.026 (0.0198) | 0.027 (0.0184)
  Basophil, Follow-up Period, n=177, 179 | 0.026 (0.0172) | 0.025 (0.0165)
  Eosinophil, Baseline Period, n=228, 231 | 0.395 (0.3292) | 0.455 (0.3859)
  Eosinophil, DB Treatment Period, n=186, 188 | 0.442 (0.3505) | 0.394 (0.3577)
  Eosinophil, Follow-up Period, n=177, 179 | 0.419 (0.3337) | 0.409 (0.3296)
  Lymphocyte, Baseline Period, n=228, 231 | 3.046 (0.9686) | 2.987 (0.9158)
  Lymphocyte, DB Treatment Period, n=177, 179 | 2.779 (0.8038) | 2.820 (0.8424)
  Lymphocyte, Follow-up Period, n=169, 173 | 2.871 (0.8784) | 2.841 (0.8107)
  WBC, Baseline Period, n=228, 231 | 7.71 (2.077) | 7.36 (1.818)
  WBC, DB Treatment Period, n=186, 188 | 7.14 (1.899) | 6.98 (1.896)
  WBC, Follow-up Period, n=177, 179 | 7.18 (1.945) | 6.96 (1.894)
  Monocyte, Baseline Period, n=228, 231 | 0.348 (0.1655) | 0.373 (0.1870)
  Monocyte, DB Treatment Period, n=186, 188 | 0.320 (0.1393) | 0.343 (0.1598)
  Monocyte, Follow-up Period, n=177, 179 | 0.334 (0.1471) | 0.326 (0.1592)
  Segmented Neu, Baseline Period, n=228, 231 | 3.892 (1.6722) | 3.517 (1.5347)
  Segmented Neu, DB Treatment Period, n=186, 188 | 3.572 (1.5407) | 3.391 (1.4828)
  Segmented Neu, Follow-up Period, n=177, 179 | 3.572 (1.5623) | 3.354 (1.4379)
  Platelet, Baseline Period, n=230, 230 | 313.8 (70.19) | 314.1 (59.46)
  Platelet, DB Treatment Period, n=187, 187 | 278.6 (55.58) | 279.5 (49.51)
  Platelet, Follow-up Period, n=175, 180 | 276.4 (49.27) | 283.6 (59.50)

9. Secondary Outcome: Mean Values for Hemoglobin
Description: Hemoglobin was assessed in participants at the indicated time points.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 231
g/L
  Baseline Period, n=231, 231 | 129.5 (7.87) | 128.4 (8.00)
  DB Treatment Period, n=186, 188 | 131.8 (7.32) | 130.8 (7.77)
  Follow-up Period, n=177, 180 | 132.1 (7.43) | 130.0 (7.90)

10. Secondary Outcome: Mean Values for Hematocrit
Description: Hematocrit was assessed in participants at indicated the time points. Hematocrit is the percentage of blood volume (BV) that is occupied by red blood cells (RBCs).
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of BV occupied by RBCs
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 231
Percentage of BV occupied by RBCs
  Baseline Period, n=231, 231 | 0.3823 (0.02296) | 0.3783 (0.02480)
  DB Treatment Period, n=186, 188 | 0.3904 (0.02291) | 0.3873 (0.02481)
  Follow-up Period, n=177, 180 | 0.3906 (0.02227) | 0.3844 (0.02416)

11. Secondary Outcome: Mean Hematology Values for Red Blood Cells (RBCs)
Description: RBCs was assessed in participants at the indicated time points.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Trillion (10^12) cells (Ti)/L
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 231 | 231
Trillion (10^12) cells (Ti)/L
  Baseline Period, n=231, 231 | 4.59 (0.312) | 4.54 (0.327)
  DB Treatment Period, n=186, 188 | 4.56 (0.303) | 4.53 (0.319)
  Follow-up Period, n=177, 180 | 4.57 (0.306) | 4.50 (0.314)

12. Secondary Outcome: Mean Values for Urine pH
Description: Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
scores on a scale
  Baseline Period, n=233, 229 | 6.02 (0.477) | 6.00 (0.536)
  DB Treatment Period, n=182, 181 | 6.02 (0.547) | 6.05 (0.507)
  Follow-up Period, n=180, 186 | 6.05 (0.538) | 6.05 (0.524)

13. Secondary Outcome: Mean Values for Urine Specific Gravity
Description: Specific gravity is a measure of the amount of material dissolved in the urine. Specific gravity is the ratio of the density (mass of a unit volume) of a substance to the density (mass of the same unit volume) of a reference substance. Normal urine has a specific gravity between 1.010 and 1.020.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
ratio
  Baseline Period, n=233, 229 | 1.0240 (0.00718) | 1.0234 (0.00673)
  DB Treatment Period, n=182, 181 | 1.0244 (0.00695) | 1.0234 (0.00649)
  Follow-up Period, n=180, 186 | 1.0237 (0.00642) | 1.0242 (0.00672)

14. Secondary Outcome: Number of Participants With the Indicated Urinalysis Results for Urine Bilirubin and Urine Nitrite
Description: Bilirubin is a normal body by-product (bile), and nitrite is a by-product of bacterial growth. Participants were categorized as Negative (Neg.) or Positive (Pos.) based on the absence or presence, respectively, of urine bilirubin (UB) and urine nitrate.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
participants
  UB-Neg, Baseline Period, n=233, 229 | 233 | 229
  UB-Pos, Baseline Period, n=233, 229 | 0 | 0
  UB-Neg, DB Treatment Period, n=182, 181 | 182 | 181
  UB-Pos, DB Treatment Period, n=182, 181 | 0 | 0
  UB-Neg, Follow-up Period, n=180, 186 | 180 | 186
  UB-Pos, Follow-up Period, n=180, 186 | 0 | 0
  Urine Nitrite-Neg, Baseline Period, n=233, 229 | 232 | 228
  Urine Nitrite-Pos, Baseline Period, n=233, 229 | 1 | 1
  Urine Nitrite-Neg, DB Treatment Period, n=182, 181 | 178 | 176
  Urine Nitrite-Pos, DB Treatment Period, n=182, 181 | 4 | 5
  Urine Nitrite-Neg, Follow-up Period, n=180, 186 | 179 | 183
  Urine Nitrite-Pos, Follow-up Period, n=180, 186 | 1 | 3

15. Secondary Outcome: Number of Participants With the Indicated Urinalysis Results for Urine Glucose, Urine Ketones, and Urine Proteins
Description: Urine glucose, urine ketones, and urine proteins were measured in participants using a dipstick (qualitative) test at the indicated time points. In this dipstick test, the level of glucose, ketones, and protein in urine samples was recorded as negative (Neg), trace (tr), 1+, 2+, and 3+ (the plus sign increases with a higher level of glucose, ketones, or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive). Participants were categorized as negative or positive based on the absence or presence, respectively, of glucose, ketones, and proteins in the urine.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
participants
  Urine Glucose-Neg, Baseline Period, n=233, 229 | 233 | 229
  Urine Glucose-Neg, DB Treatment Period, n=182, 181 | 181 | 181
  Urine Glucose-Tr, DB Treatment Period, n=182, 181 | 1 | 0
  Urine Glucose-Neg, Follow-up Period, n=180, 186 | 179 | 186
  Urine Glucose-1+, Follow-up Period, n=180, 186 | 1 | 0
  Urine Ketones-Neg, Baseline Period, n=233, 229 | 231 | 227
  Urine Ketones-Trace, Baseline Period, n=233, 229 | 0 | 1
  Urine Ketones-1+, Baseline Period, n=233, 229 | 2 | 1
  Urine Ketones-Neg, DB Treatment Period, n=182, 181 | 179 | 176
  Urine Ketones-Tr, DB Treatment Period, n=182, 181 | 3 | 5
  Urine Ketones-Neg, Follow-up Period, n=180, 186 | 180 | 184
  Urine Ketones-Trace, Follow-up Period, n=180, 186 | 0 | 1
  Urine Ketones-1+, Follow-up Period, n=180, 186 | 0 | 1
  Urine Protein-Neg, Baseline Period, n=233, 229 | 218 | 207
  Urine Protein-Trace, Baseline Period, n=233, 229 | 11 | 18
  Urine Protein-1+, Baseline Period, n=233, 229 | 2 | 4
  Urine Protein-2+, Baseline Period, n=233, 229 | 2 | 0
  Urine Protein-Neg, DB Treatment Period, n=182, 181 | 145 | 152
  Urine Protein-Tr, DB Treatment Period, n=182, 181 | 20 | 20
  Urine Protein-1+, DB Treatment Period, n=182, 181 | 14 | 7
  Urine Protein-2+, DB Treatment Period, n=182, 181 | 2 | 2
  Urine Protein-3+, DB Treatment Period, n=182, 181 | 1 | 0
  Urine Protein-Neg, Follow-up Period, n=180, 186 | 156 | 155
  Urine Protein-Trace, Follow-up Period, n=180, 186 | 16 | 22
  Urine Protein-1+, Follow-up Period, n=180, 186 | 6 | 8
  Urine Ketones-2+, Follow-up Period, n=180, 186 | 1 | 1
  Urine Ketones-3+, Follow-up Period, n=180, 186 | 1 | 0

16. Secondary Outcome: Number of Participants With the Indicated Urinalysis Results for Urine Occult Blood (OB) and the Urine Leukocyte Esterase Test (LET)
Description: Occult blood (OB) is blood that cannot be seen without a microscope. Normal urine does not contain any red blood cells. Leukocyte esterase is an enzyme and is not found in normal urine. In the dipstick (qualitative) test, the level of OB and leukocyte esterase in urine samples was recorded as negative (Neg), small, moderate, large, trace, 1+ (slightly positive), 2+ (positive), and 3+ (high positive). Participants were categorized as negative or positive based on the absence or presence, respectively, of OB and urine leukocyte esterase.
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
participants
  Urine OB-Neg, Baseline Period, n=233, 229 | 226 | 226
  Urine OB-Small, Baseline Period, n=233, 229 | 1 | 0
  Urine OB-Moderate, Baseline Period, n=233, 229 | 1 | 0
  Urine OB-Trace, Baseline Period, n=233, 229 | 4 | 3
  Urine OB-1+, Baseline Period, n=233, 229 | 1 | 0
  Urine OB-Neg, DB Treatment Period, n=182, 181 | 178 | 178
  Urine OB-Trace, DB Treatment Period, n=182, 181 | 4 | 1
  Urine OB-1+, DB Treatment Period, n=182, 181 | 0 | 1
  Urine OB-3+, DB Treatment Period, n=182, 181 | 0 | 1
  Urine OB-Neg, Follow-up Period, n=180, 186 | 177 | 184
  Urine OB-Trace, Follow-up Period, n=180, 186 | 1 | 1
  Urine OB-1+, Follow-up Period, n=180, 186 | 2 | 0
  Urine OB-2+, Follow-up Period, n=180, 186 | 0 | 1
  Urine LET-Neg, Baseline Period, n=233, 229 | 220 | 219
  Urine LET-Small, Baseline Period, n=233, 229 | 1 | 2
  Urine LET-Moderate, Baseline Period, n=233, 229 | 0 | 1
  Urine LET-Large, Baseline Period, n=233, 229 | 0 | 1
  Urine LET-Trace, Baseline Period, n=233, 229 | 7 | 0
  Urine LET-1+, Baseline Period, n=233, 229 | 3 | 2
  Urine LET-2+, Baseline Period, n=233, 229 | 0 | 2
  Urine LET-3+, Baseline Period, n=233, 229 | 2 | 2
  Urine LET-Neg, DB Treatment Period, n=182, 181 | 170 | 163
  Urine LET-Trace, DB Treatment Period, n=182, 181 | 5 | 4
  Urine LET-1+, DB Treatment Period, n=182, 181 | 5 | 6
  Urine LET-2+, DB Treatment Period, n=182, 181 | 2 | 7
  Urine LET-3+, DB Treatment Period, n=182, 181 | 0 | 1
  Urine LET-Neg, Follow-up Period, n=180, 186 | 162 | 167
  Urine LET-Trace, Follow-up Period, n=180, 186 | 5 | 5
  Urine LET-1+, Follow-up Period, n=180, 186 | 2 | 8
  Urine LET-2+, Follow-up Period, n=180, 186 | 8 | 4
  Urine LET-3+, Follow-up Period, n=180, 186 | 3 | 2

17. Secondary Outcome: Number of Participants With the Indicated Urinalysis Results for Urine Appearance (App.)/Clarity and Color
Description: Participants were assessed for their urine appearance, which was categorized as clear (normal), cloudy (presence of crystals, blood cells, or bacteria), of turbid. Also, participants were categorized by the color of urine: straw, yellow (normal urine), and dark yellow (DY) (which may be the result of bile in the urine).
Time Frame: Baseline Period (Weeks -16 to 0), DB Treatment Period (Weeks 1 to 52), and Follow-up Period (Weeks 53 to 60)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 233 | 229
participants
  Urine App.-Clear, Baseline Period, n=233, 229 | 188 | 197
  Urine App.-Cloudy, Baseline Period, n=233, 229 | 23 | 21
  Urine App.-Turbid, Baseline Period, n=233, 229 | 22 | 11
  Urine App.-Clear, DB Treatment Period, n=182, 181 | 134 | 139
  Urine App.-Cloudy, DB Treatment Period, n=182, 181 | 31 | 33
  Urine App.-Turbid, DB Treatment Period, n=182, 181 | 17 | 9
  Urine App.-Clear, Follow-up Period, n=180, 186 | 139 | 137
  Urine App.-Cloudy, Follow-up Period, n=180, 186 | 25 | 35
  Urine App.-Turbid, Follow-up Period, n=180, 186 | 16 | 14
  Urine Color-Straw, Baseline Period, n=233, 229 | 8 | 8
  Urine Color-Yellow, Baseline Period, n=233, 229 | 214 | 213
  Urine Color-DY, Baseline Period, n=233, 229 | 11 | 8
  Urine Color-Straw, DB Treatment Period, n=182, 181 | 6 | 7
  Urine Color-Yellow, DB Treatment Period, n=182,181 | 154 | 155
  Urine Color-DY, DB Treatment Period, n=182, 181 | 22 | 19
  Urine Color-Straw, Follow-up Period, n=180, 186 | 6 | 7
  Urine Color-Yellow, Follow-up Period, n=180, 186 | 156 | 160
  Urine Color-DY, Follow-up Period, n=180, 186 | 18 | 19

ADVERSE EVENTS:
Arm/Group | Placebo | FFNS 110 mcg
Serious Adverse Events (participants affected / at risk) | 4/237 | 2/237
Other Adverse Events (participants affected / at risk) | 135/237 | 129/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=237) | FFNS 110 mcg (N=237)
Appendicitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=237) | FFNS 110 mcg (N=237)
Nasopharyngitis (Infections and infestations) | 41 | 37
Bronchitis (Infections and infestations) | 24 | 34
Pharyngitis (Infections and infestations) | 18 | 12
Respiratory Tract Infection Viral (Infections and infestations) | 17 | 12
Sinusitis (Infections and infestations) | 14 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 13
Influenza (Infections and infestations) | 8 | 14
Acute Sinusitis (Infections and infestations) | 13 | 3
Tonsillitis (Infections and infestations) | 7 | 8
Gastroenteritis (Infections and infestations) | 4 | 9
Gastroenteritis Viral (Infections and infestations) | 9 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pyrexia (General disorders) | 14 | 21
Headache (Nervous system disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.